CLINICAL TRIAL: NCT00662233
Title: A Pilot Study for Soft Tissue Sarcoma
Brief Title: Combination Chemotherapy in Treating Patients With Sarcoma
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: CDR0000582271; P30CA015083 (NIH); 919110 (Other: Mayo Clinic Cancer Center); 542-91 (Other: Mayo Clinic IRB); 0791 (Registry Identifier: COGUM)
Record Dates: First submitted 2008-04-18; First posted 2008-04-21 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Ovarian Cancer; Sarcoma
Keywords: alveolar childhood rhabdomyosarcoma; previously treated childhood rhabdomyosarcoma; previously untreated childhood rhabdomyosarcoma; recurrent childhood rhabdomyosarcoma; nonmetastatic childhood soft tissue sarcoma; recurrent childhood soft tissue sarcoma; childhood desmoplastic small round cell tumor; ovarian sarcoma; stage II uterine sarcoma; stage III uterine sarcoma; embryonal childhood rhabdomyosarcoma
MeSH Terms: conditions — Ovarian Neoplasms; Sarcoma; Desmoplastic Small Round Cell Tumor | interventions — Cyclophosphamide; Doxorubicin; Etoposide; Ifosfamide; Vincristine; Chemotherapy, Adjuvant; Neoadjuvant Therapy; Brachytherapy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: etoposide
Drug: ifosfamide
Drug: vincristine sulfate
Procedure: adjuvant therapy
Procedure: neoadjuvant therapy
Procedure: therapeutic conventional surgery
Radiation: brachytherapy
Radiation: intraoperative radiation therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This clinical trial is studying how well combination chemotherapy works in treating patients with sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* To evaluate the efficacy, in terms of clinical response, pathologic response, and long-term disease-free survival, of a multidrug chemotherapy regimen patients with spindle cell or small round cell sarcoma.

OUTLINE: This is a multicenter study.

* Induction therapy: Patients receive vincristine IV, cyclophosphamide IV over 1 hour and doxorubicin hydrochloride IV over 48 hours on day 1 in week 0. Patients continue to receive vincristine IV once weekly in weeks 1 and 2. Patients also receive etoposide IV over 1 hour and ifosfamide IV over 1 hour for 5 days in week 3. Treatment repeats every 6 weeks for 2 courses.
* Local control: After completing induction therapy, patients are reevaluated for local control therapy. Some patients may undergo surgery and/or radiotherapy (e.g., brachytherapy, intraoperative radiotherapy, external beam therapy). Patients who undergo surgery begin consolidation therapy 2 weeks after completing surgery. Some patients undergo radiotherapy 5 days a week for 5½ weeks beginning at week 12 and/or after surgery (weeks 15-16).
* Consolidation therapy: Patients receive vincristine IV, doxorubicin hydrochloride IV over 1 hour, and cyclophosphamide IV over 1 hour once in weeks 12 and 18*. Patients also receive etoposide IV over 1 hour and ifosfamide IV over 1 hour for 5 days in week 15. Patients are reevaluated for local control therapy at week 21.

NOTE: *Patients undergoing radiotherapy do not receive doxorubicin hydrochloride in week 18 or week 24.

* Maintenance therapy: Patient receive vincristine IV, doxorubicin hydrochloride IV over 1 hour, and cyclophosphamide IV over 1 hour once in week 24. Patients also receive etoposide IV over 1 hour and ifosfamide IV over 1 hour for 5 days in week 21. Treatment repeats every 6 weeks for 3 courses. In week 36, patients receive vincristine, doxorubicin hydrochloride and cyclophosphamide OR etoposide and ifosfamide as before. In week 39 patients receive etoposide and ifosfamide as before.

After completion of treatment, patients are followed periodically for at least 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of any of the following:

  * High-grade nonmetastatic, nonrhabdomyosarcomatous soft tissue sarcomas (excluding undifferentiated sarcoma and Ewing sarcoma)
  * Small round cell sarcomas (excluding primitive neuroectodermal tumors of soft tissue) (closed to accrual)
  * Undifferentiated sarcomas (closed to accrual)
  * Rhabdomyosarcomas (excluding non-parameningeal head tumors, vaginal or stage I paratesticular) (closed to accrual)
  * All alveolar rhabdomyosarcomas (closed to accrual)
* No evidence distant metastatic disease (i.e., lung, bone, bone marrow)

  * Local or regional nodal disease allowed
* No spindle cell tumors of bone
* Primary lesions do not have to be resectable

PATIENT CHARACTERISTICS:

* Creatinine ≤1.5 mg/dL OR creatinine clearance > 60 mL/min/
* AST/ALT < 2 times upper limit of normal (ULN)
* Total bilirubin < 2 times ULN
* LVEF ≥ 45%
* No prior history of cancer
* Not pregnant or nursing
* Negative pregnancy test

PRIOR CONCURRENT THERAPY:

* Patients who have undergone radiation therapy after initial surgery are eligible but must have evaluation for metastatic disease within 2 weeks of starting chemotherapy
* No prior chemotherapy

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 1991-10 (Actual); Primary Completion 2013-10-21 (Actual); Study Completion 2013-10-21 (Actual)

PRIMARY OUTCOMES:
Efficacy in terms of long-term disease-free survival
Clinical response of the tumors
Pathologic response of the tumors
Long term disease-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Carola A. S. Arndt, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States